CLINICAL TRIAL: NCT01270919
Title: This Study Will be a Prospective, Non-randomized Evaluation of the Change Between Preoperative and Postoperative Outcomes for Those Who Receive the BioDuct® Device Meniscal Repair Device.
Brief Title: A Prospective, Post-market, Multi-center Feasibility Study of the BioDuct® Meniscal Repair Device
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 73
Record Dates: First submitted 2011-01-04; First posted 2011-01-05 (Estimated); Results first posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-05

CONDITIONS: Knee Meniscus Tear

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BioDuct Meniscal Repair Device (Other): BioDuct Meniscal Repair Device
  Interventions: Device: BioDuct Meniscal Repair Device

INTERVENTIONS:
Device: BioDuct Meniscal Repair Device — The BioDuct® Meniscal Repair Device is a small, cannulated, arthroscopically implanted, bioabsorbable conduit that has length sizes of 5, 7 and 9 mm. Based on the concept of trephination for treating meniscal tears in the red-white zone, the BioDuct® Meniscal Repair Device is designed to create a vascular access channel between the vascular-rich and cell-rich synovium and the meniscal tear. This channel allows for the flow of blood from the vascular to the avascular tissue to promote repair of the meniscus.
  The BioDuct® Meniscal Repair Device is not used across meniscal tears, like other fixation devices. The BioDuct® Meniscal Repair Device is used in conjunction with suturing and helps provide vascular access, while the sutures help provide fixation. Based on the Inclusion Criteria of this protocol, there can be a maximum of three BioDuct® Meniscal Repair Devices utilized for the meniscal tear.

SUMMARY:
To demonstrate repair of the meniscus at 6 months, as evaluated by MRI, will be observed; and clinical qualitative assessments will improve from preoperative to postoperative time points with the BioDuct® Meniscal Repair Device.

DETAILED DESCRIPTION:
To demonstrate repair of the meniscus 6 months postimplantation of the BioDuct® Meniscal Repair Device, utilizing MRI.

To evaluate clinical success by comparing the following qualitative criteria at 2 years postoperative to preoperative findings: effusion, swelling, pain, catching, locking, focal joint line pain and mechanical symptoms, if present preoperative. Clinical success is defined as no worsening for any of these criteria and improvement in at least one of these criteria.

ELIGIBILITY:
Inclusion Criteria:

* A. Patient has signed an IRB approved, study specific Informed Patient Consent Form.
* B. Patient is a male or non-pregnant female age 45 years or younger at time of study device implantation.
* C. Patient is a candidate for repair of one longitudinal vertical tear (bucket handle) fully located in the red-white (vascular-avascular) zone of the meniscus (3-5 mm from the synovial-meniscus junction) or repair of one longitudinal vertical tear (bucket handle) primarily located in the red-white zone of the meniscus, but partially (< 30% of total length) extending into the red zone (< 3 mm from the synovial-meniscus junction) and/or into the white zone (> 5 mm from the synovial-meniscus junction).
* D. Patient does not require more than three BioDuct® Meniscal Repair Devices for the meniscal tear.
* E. Patient requires suture only for fixation at the site where the study device will be used.
* F. Patient is willing and able to comply with postoperative scheduled MRI and clinical evaluations and rehabilitation.

Exclusion Criteria:

* G. Patient has a Body Mass Index (BMI) > 35.
* H. Patient has an active or suspected latent infection in or about the affected knee joint at time of study device implantation.
* I. Patient has horizontal, transverse, degenerative complex tears.
* J. Patient has ACL and/or PCL deficiencies within the operative knee and is not undergoing concomitant repair of these deficiencies.
* K. Patient requires bilateral meniscal repair.
* L. Patient requires meniscectomy.
* M. Patient presents with abnormal degenerative osteoarthritis of the joint [e.g. International Cartilage Repair Society (ICRS) Grade III or higher and/or Modified Outerbridge Grade III or higher].
* N. Patient has undergone previous meniscal repair to the operative knee.
* O. Patient has a knee joint with greater than 5º anatomic axis misalignment.
* P. Patient has active synovitis.
* Q. Patient is a prisoner.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2010-11; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Jack Farr, M.D., Indianapolis, Indiana
  - Jason Scopp, M.D., Salisbury, Maryland
  - Randall Holcomb, Memphis, Tennessee

RESULTS

PARTICIPANT FLOW:
Groups:
- BioDuct Meniscal Repair Device: BioDuct Meniscal Repair Device
  BioDuct Meniscal Repair Device: The BioDuct® Meniscal Repair Device is a small, cannulated, arthroscopically implanted, bioabsorbable conduit that has length sizes of 5, 7 and 9 mm. Based on the concept of trephination for treating meniscal tears in the red-white zone, the BioDuct® Meniscal Repair Device is designed to create a vascular access channel between the vascular-rich and cell-rich synovium and the meniscal tear. This channel allows for the flow of blood from the vascular to the avascular tissue to promote repair of the meniscus.
  The BioDuct® Meniscal Repair Device is not used across meniscal tears, like other fixation devices. The BioDuct® Meniscal Repair Device is used in conjunction with suturing and helps provide vascular access, while the sutures help provide fixation. Based on the Inclusion Criteria of this protocol, there can be a maximum of three BioDuct® Meniscal Repair Devices utilized for the meniscal tear.
Period: Overall Study
Arm/Group | BioDuct Meniscal Repair Device
Started | 0 (One participant was enrolled but was censored.)
Completed | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | BioDuct Meniscal Repair Device
Number analyzed (Participants) | 0
Age, Continuous [Mean (Standard Deviation); unit: years]
Sex: Female, Male [Count of Participants; unit: Participants]
Region of Enrollment [Number; unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: To Demonstrate Repair of the Meniscus 6 Months Post-implantation of the BioDuct® Meniscal Repair Device, Utilizing MRI. To Evaluate Clinical Success Using Postoperative Qualitative Criteria, as Compared to Preoperative Findings.
Time Frame: 2 years
Arm/Group | BioDuct Meniscal Repair Device
Number analyzed (Participants) | 0

2. Secondary Outcome: To Evaluate the Change in Outcomes From the Preoperative Time Point to Postoperative Time Points in Cases Implanted With the BioDuct® Meniscal Repair Device Using the SF-12, VAS Pain, WOMET and IKDC Subjective Knee Evaluation.
Time Frame: Postoperative compared to preoperative
Arm/Group | BioDuct Meniscal Repair Device
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | BioDuct Meniscal Repair Device
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other